CLINICAL TRIAL: NCT06377748
Title: The Effect of Facilitated-tucking, ShotBlocker, and the Combination of the Facilitated-tucking and ShotBlocker on Pain Caused by Hepatitis-B Vaccination in Healthy Term Infants: Randomized Controlled Study
Brief Title: The Effect of Facilitated-tucking and ShotBlocker on Pain Caused by Vaccination in Healthy Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/02
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Procedural Pain; Pain, Acute; Nursing Caries
Keywords: Healthy infant; Nonpharmacological pain management; Procedural pain
MeSH Terms: conditions — Pain, Procedural; Acute Pain | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to experimental and control groups using block randomization method. Birth weight (2500-3000 g, 3001-3500 g, 3501 g and above), gender (male and female) and mode of delivery (vaginal and cesarean section) variables will be used for block randomization.
Who Masked: Participant, Outcomes Assessor
Masking Description: Using the block randomization technique, participants will be divided into 4 groups. A web-based randomization list creation tool will be used to create the blocked randomization list. Control and intervention groups will be coded as A, B, C and D using the sealed envelope method. Randomization information will be kept from the researcher involved in data collection until data collection begins. The researcher will learn which group each baby is in just before the application (researcher blinding).
  Parents will know which group the baby is in within the scope of the research. By the nature of the sample group, babies are blind.
  Research data will be entered into the computer database by coding the group name as A, B, C and D, and statistical analysis will be performed using this coding (statistician blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Facilitated tucking position (Experimental): Newborns in this group will take the facilitated tucking position during routine Hepatitis B vaccine administration.
  Interventions: Other: Facilitated tucking position
- ShotBlocker (Experimental): ShotBlocker will be used during routine Hepatitis B vaccine administration of newborns in this group.
  Interventions: Device: ShotBlocker
- Combined facilitated tucking position and ShotBlocker (Experimental): Neonates in this group will take facilitated tucking position during routine Hepatitis B vaccine administration and ShotBlocker will be used during the procedure.
  Interventions: Combination Product: Combined facilitated tucking and ShotBlocker
- Control (No Intervention): The control group will receive routine Hepatitis B vaccination.

INTERVENTIONS:
Other: Facilitated tucking position — Neonates in this group will be given facilitated tucking position (lower and upper extremities will be held in right lateral flexion position and midline) by a volunteer nurse one minute before the vaccination procedure. The nurse will administer intramuscular vaccine injection into the vastus lateralis region of the left leg of the infant in the facilitated tucking position according to routine practice.
  Other Names: Positioning
  Arms: Facilitated tucking position
Device: ShotBlocker — Immediately prior to the vaccination procedure, the nurse will place the protruding surface of the ShotBlocker on the neonate's vaccination procedure site (left leg vastus lateralis muscle). The nurse will continue to hold the ShotBlocker at the injection site by pressing against the skin for 20 seconds. At the end of the time, she will grasp the tissue with the ShotBlocker and inject the vaccine through the opening in the center. After the procedure is completed and the needle is withdrawn, the ShotBlocker will be removed from the skin.
  Arms: ShotBlocker
Combination Product: Combined facilitated tucking and ShotBlocker — Neonates in this group will be given facilitated tucking position (lower and upper extremities will be held in right lateral flexion position and midline) by a volunteer nurse one minute before the vaccination procedure. The nurse will place the ShotBlocker on the procedure site and apply pressure to the skin for 20 seconds. At the end of the time, the nurse will grasp the tissue with the ShotBlocker and inject the vaccine through the central opening. After the injection is completed and the needle is withdrawn, the ShotBlocker will be removed from the skin. The newborn will continue to take facilitated tucking position until 1 minute after the ShotBlocker is removed.
  Arms: Combined facilitated tucking position and ShotBlocker

SUMMARY:
This study will be investigated the effects of facilitated tucking, ShotBlocker and combined facilitated tucking and ShotBlocker methods on procedural pain, crying time and duration of the procedure during Hepatitis B vaccine administration in healthy term infants.

DETAILED DESCRIPTION:
Hepatitis B vaccination is one of the painful procedures routinely performed in newborns. The pain experienced by the newborn negatively affects the prognosis of the disease, the infant's behavior, the harmony with the environment, the development of the brain and senses, as well as the family-infant interaction. Nonpharmacologic methods have been found to be effective in alleviating pain during interventions that cause pain caused by medical procedures that newborns frequently encounter. Facilitated tucking and ShotBlocker are effective methods that can be used in nonpharmacologic procedural pain management.

Studies have commonly used parent-related methods (kangaroo care, mother/father cuddling, breastfeeding, etc.) for neonatal pain management during Hepatitis B vaccine administration. In units where access to the parent is not always possible, nonpharmacologic pain methods that can be used independently of the parent can be used in the management of acute needle-related pain. In addition, no study was found in the literature comparing and combining the effect of fetal position and ShotBlocker application on hepatitis B vaccine-related pain. This study will be investigated the effects of facilitated tucking, ShotBlocker and combined facilitated tucking and ShotBlocker methods on procedural pain, crying time and duration of the procedure during Hepatitis B vaccine administration in healthy term infants.

ELIGIBILITY:
Inclusion Criteria:

* healthy term neonates
* born at 38-42 weeks gestational week,
* birth weight 2500-4400 g,
* 5th minute APGAR score above 6,
* in stable health,
* able to carry out vital activities without support,
* babies ordered Hepatitis B vaccine by the doctor

Exclusion Criteria:

* With a genetic or congenital anomaly,
* neurological, cardiological and metabolic diseases,
* in need of respiratory support,
* acute or chronic illness that causes pain,
* a complication of childbirth,
* infants of hepatitis B carrier mothers,
* nerve damage or deformity in the extremity to be vaccinated, scar tissue or incision in the vastus lateralis region,
* infants of mothers with a history of substance abuse

Ages: 38 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale | 1 min before, during, 1 min after and 3 min after the painful procedure, an average of 4-5 minutes
  The scale is used to assess procedural pain in neonates. It is a behavioral scale assessing five behavioral indicators (facial expression, cry, arms, legs, and state of alertness) and one physiological indicator (breathing patterns). Five items (facial expression, breathing pattern, arms, legs, and state of alertness) are scored as 0 (Good) or 1 (Bad), while one item (crying) is scored as 0 (Good), 1, or 2 (Bad). The total scale score ranges from 0 to 7, with higher scores indicating more pain.

SECONDARY OUTCOMES:
Crying time during the procedure | Through painful procedure completion, an average of 4 minutes
  Total crying time during the procedure is the time the newborn cries between 1 min before and 3 min after the painful procedure.
Procedure time | Through painful procedure completion, an average of 60 seconds
  For vaccine administration, it is the time between when the needle is inserted into the skin and when it is removed from the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Özdemir, PhD, Study Director — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: January through March of 2025
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Avcin E, Kucukoglu S. The Effect of Breastfeeding, Kangaroo Care, and Facilitated Tucking Positioning in Reducing the Pain During Heel Stick in Neonates. J Pediatr Nurs. 2021 Nov-Dec;61:410-416. doi: 10.1016/j.pedn.2021.10.002. Epub 2021 Oct 20. PMID 34687988
- [Background] Caglar S, Buyukyilmaz F, Cosansu G, Caglayan S. Effectiveness of ShotBlocker for Immunization Pain in Full-Term Neonates: A Randomized Controlled Trial. J Perinat Neonatal Nurs. 2017 Apr/Jun;31(2):166-171. doi: 10.1097/JPN.0000000000000256. PMID 28437308
- [Background] Drago LA, Singh SB, Douglass-Bright A, Yiadom MY, Baumann BM. Efficacy of ShotBlocker in reducing pediatric pain associated with intramuscular injections. Am J Emerg Med. 2009 Jun;27(5):536-43. doi: 10.1016/j.ajem.2008.04.011. PMID 19497458
- [Background] Kucukoglu S, Kurt S, Aytekin A. The effect of the facilitated tucking position in reducing vaccination-induced pain in newborns. Ital J Pediatr. 2015 Aug 21;41:61. doi: 10.1186/s13052-015-0168-9. PMID 26293573